CLINICAL TRIAL: NCT04167553
Title: A Phase 1, Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of HM15136(Efpegerglucagon) in Obese or Overweight Subjects With Comorbidities
Brief Title: Study for Multiple Doses of HM15136(Efpegerglucagon) in Obese or Overweight Subjects With Comorbidities
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-GCG-102
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Obese With Comorbidities; Overweight With Comorbidities; Type2 Diabetes
MeSH Terms: interventions — HM15136

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HM15136 (Experimental): HM15136 0.02mg/kg, 0.04mg/kg, 0.06mg/kg
  Interventions: Drug: HM15136
- Placebo (Placebo Comparator): Matching placebo: 0.02mg/kg, 0.04mg/kg, 0.06mg/kg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HM15136 — In Part 1, approximately 36 subjects, divided into 3 cohorts with 12 subjects (HM15136 group 9 subjects, placebo group 3 subjects) per cohort. In Part 2, approximately 66 subjects, in up to 4 cohort with 30 subjects for cohort 4 (HM15136 group 15 subjects, placebo group 15 subjects) and 12 subjects per cohorts 5-7 (HM15136 group 9 subjects, placebo group 3 subjects). Cohorts 6 and 7 are optional.
  In the end of study, Part 2 of the study consisted of 2 cohorts comprising 16 subjects total.
  Other Names: Part 1, 2
  Arms: HM15136
Drug: Placebo — In Part 1, approximately 36 subjects, divided into 3 cohorts with 12 subjects (HM15136 group 9 subjects, placebo group 3 subjects) per cohort. In Part 2, approximately 66 subjects, in up to 4 cohort with 30 subjects for cohort 4 (HM15136 group 15 subjects, placebo group 15 subjects) and 12 subjects per cohorts 5-7 (HM15136 group 9 subjects, placebo group 3 subjects). Cohorts 6 and 7 are optional.
  In the end of study, Part 2 of the study consisted of 2 cohorts comprising 16 subjects total.
  Other Names: Part 1, 2
  Arms: Placebo

SUMMARY:
The planned period of each cohort is 22 weeks including subject screening, treatments for 12 weeks, and follow up period.

DETAILED DESCRIPTION:
The current Phase I study was a two-part study. Part 1 was designed to assess the safety, PK, and pharmacodynamics (PD) after repeated doses of HM15136 in obese or overweight subjects with comorbidities (i.e., dyslipidemia and/or hypertension). Part 2 was designed to assess the safety, PK, and PD after repeated doses of HM15136 in obese or overweight subjects with T2DM and comorbidities (i.e., dyslipidemia and/or

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects
2. Age ≥ 18 to ≤ 65 years at Screening visit
3. Body Mass Index ( BMI ≥ 30 kg/m 2 or 27 kg/m 2 with presence of comorbidities (Subjects in Part 1 and Subjects with Pre diabete s mellitus (DM) in Part 2: dyslipidemia and or hypertension except for Type 2 (T2) DM, T2DM subjects in Part 2: dyslipidemia and/or hypertension with T2DM) with/without medication treatment and have had stable weight for 3 months (weight changes less than 5%)

Exclusion Criteria:

1. Previous surgical treatment for obesity (bariatric surgery, gastric banding, etc.) or any other gastrointestinal surgery that may induce malabsorption, history of bowel resection > 20 cm, any malabsorption disorder, severe gastroparesis, any GI procedure for weight loss (including LAPBAND®), as well as clinically significant gastrointestinal disorders (e.g. peptic ulcers, severe GERD ) at Screening.
2. Use of antacids, anticoagulants, or drugs that directly modify gastrointestinal (GI) motility, including antacid s anticholinergics, anticonvulsants, serotonin type 3 (5HT3) antagonists, dopamine antagonists, opiates; anticoagulation within 2 weeks of screening (But, it is not limited to the above listed drugs.)
3. Uncontrolled hypertension, defined as systolic blood pressure > 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening independent of subjects being on antihypertensive medication or no t). But, if the results are out of the reference range at the screening visit, they can be tested again on another day. Subjects with uncontrolled hypertension may be rescreened after 3 months, following initiation or adjustment of antihyp ertensive therapy.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Prosciento, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was to consist of up to 7 cohorts with a total of 102 subjects. Part 1 of the study was to consist of 3 sequential dosing cohorts, enrolling 12 subjects per cohort, for a total of 36 subjects. Part 2 of the study was to consist of up to 4 cohorts, with 30 subjects in Cohort 4 and 12 subjects per cohort for Cohorts 5-7, for a total of 66 subjects. However, during cohort 5 (0.06mg/kg) in Part 2, enrolled subjects safety data were evaluated, and decided to stop the cohort.
Pre-assignment Details: During cohort 0.06mg/kg in Part 2(cohort 5), enrolled subjects safety data were evaluated, and decided to stop the cohort. The following cohorts, cohort 6-7, were not conducted since those were optional.
Groups:
- HM15136 0.02 mg/kg Part 1: In Part 1, 0.02mg/kg cohort, there are 9 subjects.
- HM15136 0.04 mg/kg Part 1: In Part 1, 0.04mg/kg cohort, there are 9 subjects.
- HM15136 0.06 mg/kg Part 1: In Part 1, 0.06mg/kg cohort, there are 9 subjects.
- Placebo Part 1: Placebo: In Part 1, placebo cohort, there are 9 subjects.
- HM15136 0.02 mg/kg Part 2: In Part 2, 0.02mg/kg cohort 4, there are 9 subjects.
- HM15136 0.06 mg/kg Part 2: In Part 2, 0.06mg/kg cohort 5, there are 3 subjects enrollment of new subjects into Cohort 5 terminated with a lower number of subjects than planned (30).
- Placebo Part 2: In Part 2, placebo cohort, there are 4 subjects
Period: Overall Study
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
Started | 9 | 9 | 9 | 9 | 9 | 3 | 4
Completed | 8 | 9 | 6 | 7 | 6 | 1 (This cohort enrollment was discontinued after reviewing the initial safety profiles of enrolled subjects in this cohort.) | 4
Not Completed | 1 | 0 | 3 | 2 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: During Part 2 0.06mg/kg(cohort 5), the safety profile of enrolled subjects were evaluated, and decided to stop enrolling subjects. Planned cohorts, cohort 6 to 7, were not conducted since those were optional.
Groups:
- HM15136 0.02 mg/kg Part 1: HM15136: In Part 1, approximately 36 subjects, divided into 3 cohorts with 12 subjects (HM15136 group 9 subjects, placebo group 3 subjects) per cohort.
- HM15136 0.04 mg/kg Part 1: HM15136 0.04 mg/kg
  HM15136: In Part 1, approximately 36 subjects, divided into 3 cohorts with 12 subjects (HM15136 group 9 subjects, placebo group 3 subjects) per cohort.
- HM15136 0.06 mg/kg Part 1: HM15136 0.06 mg/kg
  HM15136: In Part 1, approximately 36 subjects, divided into 3 cohorts with 12 subjects (HM15136 group 9 subjects, placebo group 3 subjects) per cohort.
- Placebo Part 1: Placebo: In Part 1, approximately 36 subjects, divided into 3 cohorts with 12 subjects (HM15136 group 9 subjects, placebo group 3 subjects) per cohort.
- HM15136 0.02 mg/kg Part 2; Placebo Part 2: In Part 2, approximately 66 subjects, in up to 4 cohort with 30 subjects for cohort 4 (HM15136 group 15 subjects, placebo group 15 subjects) and 12 subjects per cohorts 5-7 (HM15136 group 9 subjects, placebo group 3 subjects). Cohorts 6 and 7 are optional.
- HM15136 0.06 mg/kg Part 2: HM15136 0.06 mg/kg Part 2
  In Part 2, approximately 66 subjects, in up to 4 cohort with 30 subjects for cohort 4 (HM15136 group 15 subjects, placebo group 15 subjects) and 12 subjects per cohorts 5-7 (HM15136 group 9 subjects, placebo group 3 subjects). Cohorts 6 and 7 are optional.
- Total: Total of all reporting groups
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2 | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 3 | 4 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 9 | 3 | 4 | 52
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 4 | 4 | 6 | 1 | 0 | 25
  Male | 2 | 6 | 5 | 5 | 3 | 2 | 4 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 1 | 1 | 0 | 0 | 7
  White | 8 | 7 | 6 | 6 | 8 | 3 | 4 | 42
  More than one race | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 9 | 3 | 4 | 52

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Incidence of AEs
Description: To evaluate the incidence of AEs: Skin and subcutaneous tissue disorders
Time Frame: after multiple subcutaneous (SC) doses for 12 weeks
Population: To evaluate Skin and subcutaneous tissue disorders occurance from baseline to end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 6 | 2 | 4
Participants | 1 | 2 | 4 | 2 | 2 | 0 | 3

2. Primary Outcome: To Evaluate Serum Amylase Levels at 12 Weeks
Description: To evaluate the incidence of clinical lab abnormalities of serum amylase
Time Frame: after multiple subcutaneous (SC) doses for 12 weeks
Population: incidence of clinical lab abnormalities comparing from baseline to end of treatment
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- HM15136 0.02 mg/kg Part 2: In Part 2, 0.02mg/kg cohort, there are 9 subjects
- HM15136 0.06 mg/kg Part 2: In Part 2, 0.06mg/kg cohort, there are 15 subjects
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
Number analyzed (Participants) | 8 | 9 | 6 | 7 | 6 | 1 | 4
U/L | 0.1 (12.17) | -1.1 (8.13) | 7.8 (8.93) | -3.6 (8.18) | -12.5 (50.69) | -2 (NA) — n=1 so there was no SD | -11 (15.21)

3. Primary Outcome: Change From Baseline in Tympanic Temperature
Description: tympanic temperature change
Time Frame: after multiple subcutaneous (SC) doses for 12 weeks
Population: Evaluation of body temperature from baseline to end or treatment
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 1 | 4
Celsius | -0.28 (0.471) | -0.08 (0.291) | -0.23 (0.372) | -0.10 (0.408) | -0.1 (0.533) | -0.1 (NA) — n=1 so there was no SD | -0.03 (0.411)

4. Primary Outcome: Change From Baseline in 12-lead ECG Parameters
Description: QT interval corrected for HR using Fridericia's correction [QTcF]
Time Frame: after multiple subcutaneous (SC) doses for 12 weeks
Population: To evaluate 12-lead ECG parameters changes from baseline to end of treatment
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 6 | 1 | 4
msec | -26.6 (22.40) | -13.5 (14.98) | 20.5 (10.14) | -13.2 (14.02) | -10 (18.24) | 10.3 (NA) — N=1, so there was no SD | 14.0 (10.85)

5. Primary Outcome: Injection Site Reactions
Description: Injection site reactions occurance
Time Frame: after multiple subcutaneous (SC) doses for 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 3 | 4
Participants | 1 | 3 | 2 | 0 | 1 | 0 | 1

6. Secondary Outcome: Serum Lipid Profiles
Description: Change Cholesterol from baseline to end of treatment (12 weeks)
Time Frame: Change from baseline to end of treatment (12 weeks)
Population: Change Cholesterol from baseline to end of treatment
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 6 | 1 | 4
mg/dL | -4.94 (3.71) | 1.15 (3.68) | 2.56 (4.07) | -3.69 (3.94) | -7.41 (19.01) | 30.52 (NA) — n=1 so there is no SE | -0.25 (8.79)

ADVERSE EVENTS:
Time Frame: Screening, week 1, week 3, week 5, week 9, week 13, week 17
Arm/Group | HM15136 0.02 mg/kg Part 1 | HM15136 0.04 mg/kg Part 1 | HM15136 0.06 mg/kg Part 1 | Placebo Part 1 | HM15136 0.02 mg/kg Part 2 | HM15136 0.06 mg/kg Part 2 | Placebo Part 2
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/9 | 2/9 | 4/9 | 2/9 | 2/9 | 0/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HM15136 0.02 mg/kg Part 1 (N=9) | HM15136 0.04 mg/kg Part 1 (N=9) | HM15136 0.06 mg/kg Part 1 (N=9) | Placebo Part 1 (N=9) | HM15136 0.02 mg/kg Part 2 (N=9) | HM15136 0.06 mg/kg Part 2 (N=3) | Placebo Part 2 (N=4)
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 2 | 2 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT04167553/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT04167553/SAP_001.pdf